

Appendix No. 1 to Appendix No. 1 to Regulations of the Bioethics Committee at ICZMP introduced by Order No. 36/2022 of the Director of ICZMP of 16/05/2022

## INFORMED CONSENT OF THE PATIENT AND/OR STATUTORY REPRESENTATIVES TO PARTICIPATE IN A MEDICAL EXPERIMENT AND PROCESSING OF PERSONAL DATA

**Title of the medical experiment/research:** The use of MET-PET combined with MRI in surgical treatment and postoperative radiotherapy of glioblastoma multiforme - a randomized, blinded, prospective study.

Details of the person referred for testing: Name: Last name: PESEL: In the case of a person who does not have a PESEL number - name and number of another document confirming identity: Details of the parent or legal guardian (complete if the person referred for testing is a minor): Name: Last name: PESEL: In the case of a person who does not have a PESEL number - name and number of another document confirming identity: Data of the second parent or legal guardian (complete if the person referred for examination is a minor): Name: Last name: PESEL: *In the case of a person who does not have a PESEL* number - name and number of another document confirming identity:

(In the case of minor Participants, it is necessary to express written consent from each of the legal representatives of the minor and their joint consent and:

- for Participants who are under 13 years of age signed by the child's parents/legal representatives and the child himself, if he is able to understand the information regarding

Informed consent form for participation in a medical experiment and processing of personal data version of May 16, 2022 page 1



the examination being conducted. If a child does not consent to the proposed study, he or she cannot participate in the study.

- for Participants who are over 13 years of age and they are under 18 years of age , signed by Participants and parents/legal representatives of the child)

| I | declare | that | I | have | been | informed | (a) |
|---|---|---|---|---|---|---|---|
| | nd threats, any i | | | | | expected benefity, and about my | |
| | | | | | | rmation form reg<br>y answers to the | |
| I was in | nformed that part | cicipation in t | he medical | experiment is v | oluntary. | | |
| without<br>conseque<br>further | giving a reason<br>nences in the form | n. I have been of any discretized in a new discreti | n informed<br>rimination,<br>ave receive | that exercising including the ri | g this right we ght to health | draw consent) at will have no neg care, and will no of this form and | ative legal<br>t affect the |
| a fragn | | rative materi | ial taken a | s part of medi- | | ogical material (w<br>t/procedure, othe | |
| conduct<br>by | ting the study | in accordan | ce with p | olicy no | | caused in connection offor paying comparing | issued |
| _ | e my full, i<br>nent/research. | nformed a | nd volun | tary consent | to partic | cipate in this | medical |
| Patient: | | | | | | | |
| (name a | and surname) | (sign | nature) | | (da | te) | |
| Parent | /legal guardian: | | | | | | |
| (name a | and surname) | (sign | nature) | | (da | te) | ••• |
| II Pare | nt/legal guardia | an: | | | | | |
| (name a | and surname) | (sign | nature) | | (da | te) | |

Informed consent form for participation in a medical experiment and processing of personal data version of May 16, 2022 page 2



I, the undersigned, declare that I have explained to the Patient the details of the proposed examination, as described in the patient information form. Before any procedures were undertaken, I discussed with the Patient his/her participation in the entire research program, informing about the goals and nature of the clinical trial as well as the benefits and risks resulting from participation in this study. When talking to the patient, I discussed the presented study using understandable, possibly simple terms and provided explanations regarding the essence and importance of the study.

| Person obtaining consent for the s | study: | |
|------------------------------------|-------------|--------|
| (name and surname) | (signature) | (date) |



## INFORMED CONSENT OF THE PATIENT AND/OR STATUTORY REPRESENTATIVES TO THE PROCESSING OF PERSONAL DATA

Title of the medical experiment/research:

The use of MET-PET combined with MRI in surgical treatment and postoperative radiotherapy of glioblastoma multiforme - a randomized, blinded, prospective study.

## I consent to the processing of my data

data in this study in accordance with the law in force in Poland (Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 on the protection of natural persons with regard to the processing of personal data and on the free movement of such data and repealing Directive 95 /46/EC). I consent to the transfer of my anonymous data to other countries, both within and outside Europe. However, the data analyzed by the relevant authorities, representatives of the Ministry of Health, the study sponsor and its representatives, the US Food and Drug Administration (FDA) and other government organizations and bioethics committees will be available only in anonymous form.

## I have been informed that:

Dationt:

- a. the data controller is the Provincial Multidisciplinary Center of Oncology and Traumatology.
  M. Kopernika in Łódź ( WWCOiT ), ul. Pabianicka 62, 93-513 Łódź
- b. The Data Protection Inspector at WWCOiT is Mr. Tomasz Zdzienicki, e-mail <a href="mailto:iod@kopernik.lodz.pl">iod@kopernik.lodz.pl</a> My personal data will be processed for the purpose of carrying out the study Application of MET-PET combined with MRI in the surgical treatment and postoperative radiotherapy of glioblastoma multiforme a randomized, blinded, prospective study.
- c. in WWCOiT pursuant to Art. 9 section 2 letter a of the general regulation on the protection of personal data of April 27, 2016.
- d. about the method of data processing, the right to access them, submit an application for rectification, deletion, limitation of processing, and the right to lodge a complaint with the Personal Data Protection Office.

I have been informed that if I withdraw my consent to participate in the study, the data collected so far may be used and processed as part of the study database.

| rationt. | | |
|---------------------------|-------------|--------|
| (name and surname) | (signature) | (date) |
| I Parent/legal guardian: | | |
| (name and surname) | (signature) | (date) |
| II Parent/legal guardian: | | |
| (name and surname) | (signature) | (date) |

Informed consent form for participation in a medical experiment and processing of personal data version of May 16, 2022 page 4